CLINICAL TRIAL: NCT00790556
Title: A Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK8245.
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK8245 (8245-004)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8245-004; 2008_582
Record Dates: First submitted 2008-11-07; First posted 2008-11-13 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (5-(3-(4-(2-bromo-5-fluorophenoxy)piperidin-1-yl)isoxazol-5-yl)-2H-tetrazol-2-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK8245
  Interventions: Drug: MK8245
- 2 (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK8245 — MK8245 50 mg capsules twice daily for 13 days. On Day 14, only the morning dose of study medication will be taken. There will be a 14 day washout period. Patients will then crossover to MK8245 placebo capsules twice daily for 13 days. On Day 14, only the morning dose of study drug will be taken.
  Arms: 1
Drug: Comparator: Placebo — MK8245 placebo capsules twice daily for 13 days. On Day 14, only the morning dose of study medication will be taken. There will be a 14 day washout period. Patients will then crossover to MK8245 50 mg capsules twice daily for 13 days. On Day 14, only the morning dose of study drug will be taken.
  Arms: 2

SUMMARY:
A 2-period crossover study to assess the safety, tolerability and glucose-lowering effects of MK8245.

DETAILED DESCRIPTION:
Hypothesis: Multiple doses of MK-8245 are sufficiently safe and well tolerated in patients with Type 2 diabetes based on an assessment of clinical and laboratory adverse experiences (AEs), to permit continued clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of Type 2 Diabetes and is being treated with diet and exercise alone or a single oral anti-hyperglycemic agent
* Subject is willing to follow the weight-maintaining diet and exercise program or equivalent beginning 4 weeks before receiving study drug, throughout the study and until the post study visit
* Subject has been a nonsmoker and/or has not used nicotine-containing products for at least approximately 6 months

Exclusion Criteria:

* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of neoplastic disease (except non-melanomatous skin carcinoma, carcinoma in situ of the cervix, other malignancies successfully treated at least 10 years prior to screening, or malignancies deemed highly unlikely to recur.)
* Subject has a history of Type 1 Diabetes Mellitus and/or history of ketoacidosis
* Subject has a history of contact lens use within approximately the previous 6 months
* Subject has been diagnosed with dry eye syndrome
* Subject has used lipid-lowering therapies in the past 3 months (Subjects on a stable monotherapy dose of statins may be included)
* Subject has had major surgery, donated or lost 1 unit of blood or participated in another investigational study within 4 weeks of starting in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Nio Y, Hasegawa H, Okamura H, Miyayama Y, Akahori Y, Hijikata M. Liver-specific mono-unsaturated fatty acid synthase-1 inhibitor for anti-hepatitis C treatment. Antiviral Res. 2016 Aug;132:262-7. doi: 10.1016/j.antiviral.2016.07.003. Epub 2016 Jul 5. PMID 27392483

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For subjects taking anti-hyperglycemic agents and who otherwise qualified for the study, a 4-week washout/run-in period was required prior to dosing.
Groups:
- MK8245 Then Placebo: During Treatment Period 1, these subjects received MK-8245 50 mg twice daily 12 hours apart for 13 days, only the AM dose was administered on Day 14.
  During Treatment Period 2, these subjects received MK-8245 matching placebo twice daily 12 hours apart for 13 days, only the AM dose was administered on Day 14.
- Placebo Then MK8245: During Treatment Period 1, these subjects received MK-8245 matching placebo twice daily 12 hours apart for 13 days, only the AM dose was administered on Day 14.
  During Treatment Period 2, these subjects received MK-8245 50 mg twice daily 12 hours apart for 13 days, only the AM dose was administered on Day 14.
Period: Treatment Period 1
Arm/Group | MK8245 Then Placebo | Placebo Then MK8245
Started | 8 | 6
Completed | 6 | 6
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout After Period 1
Arm/Group | MK8245 Then Placebo | Placebo Then MK8245
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | MK8245 Then Placebo | Placebo Then MK8245
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 49.43 [30 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinical and Laboratory Adverse Events (CAEs and LAEs)
Description: An LAE is defined as any unfavorable & unintended change in the chemistry of the body temporally associated with the use of study product, whether or not considered related to the use of the product. A CAE is defined similarly but also includes changes in structure or function of the body.
  Serious AEs are those occuring that result in one or more of the pre-specified outcome(s) that meet the criteria of seriousness, including death, life-threatening, significant disability, or hospitalization, etc.
  Drug-relatedness was determined by the investigator based on clinical judgement.
Time Frame: 56 days
Population: All 14 subjects enrolled in the study were included in the assessment of safety and tolerability (although only 12 subjects received placebo, our database includes all subjects in the analysis).
Measure: Number; unit: participants
Groups:
- MK8245: MK-8245 50 mg twice daily 12 hours apart for 13 days, only the AM dose was administered on Day 14.
  Includes results of this treatment from both treatment periods.
- Placebo: MK-8245 matching placebo twice daily 12 hours apart for 13 days, only the AM dose was administered on Day 14.
  Includes results of this treatment from both treatment periods.
Arm/Group | MK8245 | Placebo
Number analyzed (Participants) | 14 | 14
participants
  With clinical adverse events (CAEs) | 4 | 5
  With drug-related CAEs | 0 | 0
  With Serious CAEs | 0 | 0
  With laboratory adverse events (LAEs) | 0 | 0
  With drug-related LAEs | 0 | 0
  With serious LAEs | 0 | 0

2. Primary Outcome: Mean Change From Baseline in Hepatic Glucose Production (HGP) at Day 14
Description: Changes in HGP were determined during a euglycemic clamp procedure. HGP was evaluated as milligrams per kilogram of glucose produced per minute.
Time Frame: Day 14 of each 14-day Treatment Period
Population: Subjects who discontinued were not used in the analysis.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | MK8245 | Placebo
Number analyzed (Participants) | 12 | 12
mg/kg/min | -1.09 (1.54) | -0.87 (0.94)

3. Other Pre Specified Outcome: Hepatic Glucose Production (HGP) at Baseline
Time Frame: Baseline
Population: Subjects who discontinued were not used in the analysis.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | MK8245 | Placebo
Number analyzed (Participants) | 12 | 12
mg/kg/min | 1.87 (0.36) | 1.95 (0.36)

ADVERSE EVENTS:
Time Frame: Treatment Period 1, Days 1 to 14, 14 day washout, Treatment Period 2, Days 1 to 14, 14 days to post study.
Description: Spontaneous collection of all AEs; All 14 subjects enrolled in the study were included in the assessment of safety and tolerability (although only 12 subjects received placebo, our database includes all subjects in the analysis).
Arm/Group | MK8245 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 4/14 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK8245 (N=14) | Placebo (N=14)
Cataract (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Infusion site haemorrhage (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Body tinea (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Stat. analysis of HGP was not performed as insulin suppression lead to a near complete suppression of HGP in both placebo and MK-8245 treated subjects, making it impossible to determine if MK-8245 could lead to a greater insulin effect than placebo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.